CLINICAL TRIAL: NCT05559242
Title: To Evaluate the Phase I Pharmacokinetics of Anlotinib Hydrochloride Capsules in Liver Dysfunction Patients and Healthy Subjects
Brief Title: Pharmacokinetic Study of Anlotinib Hydrochloride Capsules in Healthy Subjects and Liver Dysfunction Patients
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ALTN-I-10
Record Dates: First submitted 2022-09-27; First posted 2022-09-29 (Actual); Last update posted 2022-09-29 (Actual); Status verified 2022-09

CONDITIONS: Liver Dysfunction
MeSH Terms: conditions — Liver Diseases

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Anlotinib Hydrochloride Capsules (Experimental): Anlotinib hydrochloride capsules, 12mg, 1 time in total
  Interventions: Drug: Anlotinib Hydrochloride Capsule

INTERVENTIONS:
Drug: Anlotinib Hydrochloride Capsule — Anlotinib hydrochloride is a muti-target tyrosine kinase inhibitor

SUMMARY:
To evaluate the pharmacokinetic difference of anlotinib hydrochloride capsule between mild/moderate liver dysfunction subjects and healthy subjects, and to provide basis for formulating the clinical drug regimen for patients with liver dysfunction.

ELIGIBILITY:
Inclusion Criteria:

* Criteria 1 to 4 are applicable to all subjects.

  1. The subjects volunteered to participate in the study, signed the informed consent, and had good compliance;
  2. Age: 18-75 years old (including both end values) (the healthy subject group and the liver dysfunction group are age matched, the mean is ± 10 years); Both male and female (healthy subjects group and liver dysfunction group were matched by gender, mean ± 1 case);
  3. Body mass index (BMI) ≥ 18 and ≤ 30 kg / m2, and male weight ≥ 50 kg or female weight ≥ 45 kg (weight matching between healthy subjects and liver dysfunction group, mean ± 10%);
  4. Female subjects of childbearing age should agree to use contraceptive measures (such as IUDs, contraceptives or condoms) during the study and within 6 months after the end of the study; Serum pregnancy test was negative within 7 days before study enrollment, and must be a non lactating subject; Male subjects should agree to use contraceptives during the study period and within 6 months after the end of the study period;
* Criteria 5 to 8 are applicable to subjects with liver dysfunction. 5. For the subjects with liver dysfunction, they are diagnosed as chronic (≥ 6 months) stable liver function impairment through past medical history, physical examination, serological indicators (such as albumin, bilirubin, glutamic pyruvic transaminase, glutamic oxaloacetic transaminase, prothrombin time, etc.), liver biopsy or imaging (such as computed tomography, magnetic resonance imaging, ultrasound, laparoscopy, etc.); 6. Subjects with liver dysfunction caused by previous primary liver diseases and assessed as grade A / mild (5-6 points) or grade B / moderate (7-9 points) according to child Pugh grading score (albumin was not used within 14 days); 7. The main organs have good functions and meet the following standards: The blood routine examination shall meet the following standards (no blood transfusion or correction with hematopoietic stimulator drugs within 7 days before screening): hemoglobin (Hgb) ≥ 90g / L; Neutrophil absolute value (neut) ≥ 1.5 × 109/L; Biochemical examination shall meet the following standards: serum creatinine (CR) ≤ 1.5 × ULN or creatinine clearance rate (CCR) ≥ 60ml / min; Liver function test shall meet the following standards: alanine transferase (ALT) and aspartate transferase (AST) ≤ 5 × ULN; Coagulation function test shall meet the following standards: prothrombin time (PT) extension ≤ 6S, prothrombin activity (PTA) ≥ 40%; Cardiac color Doppler evaluation: left ventricular ejection fraction (LVEF) ≥ 50%; 8. No drugs affecting CYP3A4 were used within 2 weeks before the study;
* Criteria 9, 10 are applicable to healthy subjects. 9. Main organ function is good, laboratory examination (blood routine, blood biochemistry, coagulation function, etc.), cardiac color ultrasound, 12 lead electrocardiogram, abdominal B-ultrasound and other examinations are normal or abnormal, but they are judged by the investigator to be of no clinical significance; 10. Those who did not use any prescription drugs, over-the-counter drugs, Chinese herbal medicines or food supplements within 2 weeks before the study medication;

Exclusion Criteria:

* Exclusion criteria 1 to 15 are applicable to all subjects.

  1. Allergic constitution, including severe drug allergy or drug allergy history; Those who are known to be allergic to anlotinib hydrochloride capsules or their excipients;
  2. Those who lost blood or donated blood ≥ 450 ml or received blood transfusion within one month before screening; Or having taken any clinical trial drug;
  3. Alcohol breath test is positive or there is a history of alcoholism within 2 weeks before screening (drinking 14 units of alcohol per week: 1 unit = 360ml of beer or 45ml of spirits with 40% alcohol or 150ml of wine); Those who cannot abstain from smoking and drinking during the test;
  4. Those with serious infection, trauma, gastrointestinal surgery or other major surgical operations within 4 weeks before screening;
  5. There are many factors that affect oral administration and drug absorption (such as inability to swallow, gastrointestinal tract resection, ulcerative colitis, symptomatic / inflammatory bowel disease, chronic diarrhea, intestinal obstruction and other digestive tract diseases);
  6. Those who have taken in special diet (such as grapefruit juice / grapefruit juice, methyl xanthine rich coffee, tea, cola, chocolate, energy drinks, etc.) or have taken strenuous exercise or other factors affecting drug absorption, distribution, metabolism, excretion, etc. within 2 days before the study medication;
  7. Those with a history of drug abuse or positive drug screening;
  8. Those who have taken the study drug or participated in clinical trials of other drugs and taken the study drug within one month before screening;
  9. Female subjects who are breastfeeding or whose serum pregnancy results are positive during the screening period;
  10. Have a history of malignant tumor in the past 5 years (except for cured skin basal cell carcinoma and cervical carcinoma in situ);
  11. HIV antibody positive;
  12. There are any serious and / or uncontrollable diseases, including:

      1. blood pressure control is not ideal (systolic blood pressure ≥ 150mmhg or diastolic blood pressure ≥ 100 mmHg);
      2. Have grade ≥ 2 myocardial ischemia or myocardial infarction, arrhythmia (including QTc ≥ 480ms) and grade ≥ 2 congestive heart failure;
      3. Arterial / venous thrombosis events occurred within 6 months, such as cerebrovascular accidents (including transient ischemic attack, cerebral hemorrhage, cerebral infarction), deep vein thrombosis and pulmonary embolism;
  13. There are other serious physical or mental diseases, or the history and / or abnormal clinical laboratory tests that the investigator considers may affect the test results, including but not limited to the history of circulatory system, endocrine system, nervous system, digestive system, urinary system or blood, immune, mental and metabolic diseases (excluding the primary liver diseases of patients with liver dysfunction);
  14. There is a history of live attenuated vaccine vaccination within 2 weeks before screening or live attenuated vaccine vaccination is planned during the trial;
  15. According to the judgment of the investigator, there are concomitant diseases that seriously endanger the safety of the subject or affect the completion of the study, or subjects who are considered unsuitable for enrollment for other reasons;
* Exclusion criteria 16 is only applicable to subjects with liver dysfunction 16. Subjects with liver dysfunction can not be included in the group if they have any of the following conditions:

  1. drug-induced liver injury;
  2. Liver transplantation;
  3. Patients with acute liver function injury caused by various reasons within 2 months before screening;
  4. Patients with severe peritoneal effusion or pleural effusion requiring puncture drainage;
  5. Patients with hepatorenal syndrome;
  6. Patients with biliary cirrhosis, biliary obstruction, cholestatic liver disease and other diseases affecting bile excretion;
  7. Patients with severe portal hypertension or who have received previous portosystemic shunt, including transjugular intrahepatic portosystemic shunt;
  8. Patients in the state of liver failure at present, or patients with cirrhosis complicated with obvious hepatic encephalopathy, liver cancer, rupture and bleeding of esophageal and gastric varices and other complications that researchers think are inappropriate;
* Exclusion criteria 17 is only applicable to healthy subjects. 17. Hepatitis B surface antigen (HBsAg) positive or HCV-RNA positive.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-10 (Estimated); Primary Completion 2023-06 (Estimated); Study Completion 2023-07 (Estimated)

PRIMARY OUTCOMES:
Peak concentration (Cmax) | predose, 1,2,4,8,11,24,48,96,144,192,240,336 hours after administration
  Maximum plasma drug concentration
Area under curve (0-t) | predose, 1,2,4,8,11,24,48,96,144,192,240,336 hours after administration
  Area under the plasma concentration-time curve from time 0 to last time of quantifiable concentration
Area under curve (0-∞) | predose, 1,2,4,8,11,24,48,96,144,192,240,336 hours after administration
  Area under the plasma concentration-time curve from time 0 and extrapolated to infinite time

SECONDARY OUTCOMES:
Time to reach maximum concentration (TMAX) | predose, 1,2,4,8,11,24,48,96,144,192,240,336,hours after administration
  Time to reach maximum concentration (TMAX)
Elimination half life (t1/2) | predose, 1,2,4,8,11,24,48,96,144,192,240,336,hours after administration
  Elimination half life (t1/2)
Apparent clearance (CL/F) | predose, 1,2,4,8,11,24,48,96,144,192,240,336,hours after administration
  Apparent clearance (CL/F)
Apparent distribution volume (Vd/F) | predose, 1,2,4,8,11,24,48,96,144,192,240,336,hours after administration
  Apparent distribution volume (Vd/F)
Adverse event rate | From the first administration to 15 days after the administration
  Incidence and severity of adverse events and serious adverse events, and abnormal laboratory examination indicators

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - The Second Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - Hunan Cancer Hospital, Changsha, Hunan

IPD SHARING:
Plan to Share IPD: No